CLINICAL TRIAL: NCT02452073
Title: An Analysis of the Relative Risk for Low Triiodothyronine Syndrome in Patients With Chronic Radiation Enteritis
Status: Completed | Type: Observational
Sponsor: Shengxian Fan (Other)
Responsible Party: Sponsor-Investigator, Shengxian Fan, M.D., Jinling Hospital, China
Organization: Jinling Hospital, China (Other)
Other Study IDs: JinlingH
Record Dates: First submitted 2015-05-15; First posted 2015-05-22 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: The Clinical Incidence of Low Triiodothyronine Syndrome
Keywords: low triiodothyronine syndrome; chronic radiation enteritis; triiodothyronine; thyroxine; thyroid stimulating hormone
MeSH Terms: conditions — Euthyroid Sick Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- CRE group: patients with chronic radiation enteritis
  Interventions: Other: Thyroid function tests
- malignancy group: patients with some kinds of malignant tumors but had not previously received radiotherapy
  Interventions: Other: Thyroid function tests
- control group: age-matched healthy volunteers
  Interventions: Other: Thyroid function tests

INTERVENTIONS:
Other: Thyroid function tests

SUMMARY:
Radiation enteritis (RE) is by simple definition an inflammatory process occurring at the level of the intestines as a response to abdominal or pelvic radiation energy exposure. Due to the dosage of radiation, sensitivity of organs to radiation, and some patient characteristics, RE can present as either an acute or chronic syndrome. Clinical manifestations differ but may include abdominal pain, malabsorption, diarrhea, cachexia, intestinal bleeding, obstruction, and even perforation, which compromise quality of life. For many years, radiotherapy of the abdominal or pelvic region is commonly used for a significant percentage of patients with rectosigmoid and genitourinary system tumors. Different techniques have been developed to prevent the occurrence of radiation induced injury. However, the incidence of CRE is expected to continue to rise during the coming years. What's more, abdominal or pelvic radiotherapy can also lead to other side effects in addition to RE, such as skin desquamation, local soft tissue injury, and so on. Till now, lots of attention is only paid to local complications, there is little report on systemic damage of abdominal or pelvic radiotherapy.

Low triiodothyronine syndrome (LT3S), a condition characterized by low circulating triiodothyronine (T3) levels, normal thyroxine (T4), free thyroxine (FT4) and thyroid-stimulating hormone (TSH) levels in the absence of an intrinsic thyroid disease, is variously known as the "nonthyroidal illness syndrome (NTIS)". This condition is frequently detected in critical illness. Reichlin et al. first noticed that some aspects of thyroid hormone metabolism might change during many chronic illnesses as early as 1973. Data has shown that about 35-70% of acute and chronic critical conditions were associated with a significant abnormal thyroid hormone metabolism, of which LT3S was the most common type. Furthermore, these changes have been shown to be associated with disease severity and have been connected with poor short-term prognosis.

To date, there are lots of literatures include detailed reports on the relationship between LT3S and chronic illnesses such as rheumatoid arthritis, systemic lupus erythematosus, sepsis, and so on. However, no systematic analysis of LT3S in patients with CRE has been undertaken. As such, the present study aimed to investigate the frequency of LT3S in CRE patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic radiation enteritis
* patients with some kinds of malignant tumors but had not previously received radiotherapy
* age-matched healthy volunteers

Exclusion Criteria:

* Patients with a chronic disease other than CRE, including RA, SLE, thyroid illness, infectious diseases, and hepatic or renal disorders were excluded.
* patients have taken any drugs that may influence thyroid hormone secretion and metabolism during the previous 3 months.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients and volunteers who were admitted to our hospital
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
morbidity | one year
  The results will be expressed as percentage